CLINICAL TRIAL: NCT06747403
Title: The Sensitivity, Specificity and Predictive Accuracy of Gastric Point of Care Ultrasound in Pediatric Trauma Patients
Brief Title: Accuracy of Gastric POCUS in Pediatric Trauma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor, Assiut University
Other Study IDs: Gastric Pocus
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Trauma Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to detect the predictive accuracy of the gastric POCUS in pediatric trauma patients undergoing urgent and semi urgent operative procedures.

The main question it aims to answer is :

What is the predictive value of the gastric POCUS in pediatric patients? Participants are pediatric patients who will be scheduled for operative procedures within one hour of performing gastric POCUS.

DETAILED DESCRIPTION:
Reflux aspiration of gastric contents is a critical concern in the perioperative setting, as it can result in severe complications such as aspiration pneumonia, acute respiratory distress syndrome, and even death. The risk is heightened during general anesthesia and is influenced by the quality and quantity of stomach contents. To mitigate this risk, the American Society of Anesthesiologists (ASA) recommends fasting guidelines prior to elective procedures. However, factors like trauma, acute and chronic pain, opioid use, and certain medical conditions can delay gastric emptying, complicating adherence to these guidelines.

Recent advancements in ultrasound techniques enable comprehensive evaluations of the nature and volume of gastric contents, making this tool convenient, noninvasive, and applicable at the bedside with minimal contraindications.The Perlas Model has been developed to identify surgical patients with "at-risk" stomachs, aiding in preoperative planning and airway management during general anesthesia. This model facilitates decisions regarding rapid sequence induction (RSI) and the choice of airway management techniques. However, there is a notable lack of research focusing on the use of ultrasound techniques in pediatric trauma patients to determine their diagnostic performance and predictive accuracy regarding gastric contents. Therefore, the aim of this study is to investigate the efficacy of POCUS in assessing the nature and volume of gastric contents in pediatric trauma patients undergoing urgent and semi-urgent surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients who will be scheduled for operative procedures within an hour of performing gastric POCUS.
2. Age group 1-18 years
3. ASA Physical status (I-III).
4. Both gender

Exclusion Criteria:

1. Children with known abnormal upper GIT anatomy or prior upper GIT surgery.
2. Children with wounds of the epigastrium precluding probe placement.
3. Children deemed unable to tolerate the US probe

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: This study will be conducted in the emergency departments in Assiut and Suez Canal University hospitals after its approval from the ethical committees.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of gastric POCUS | 1 hour from performing gastric POCUS till performing operative procedures
  We will investigate the diagnostic performance and predictive accuracy of the gastric POCUS in pediatric trauma patients undergoing urgent and semi urgent operative procedures as our primary outcome of interest. The sensitivity, specificity, positive predictive value and negative predictive value will be assessed using the Receiver Operating Characteristics (ROC) curve.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No